CLINICAL TRIAL: NCT05112705
Title: Diagnosing Deep-vein Thrombosis Early in Critically Ill Patients (DETECT) Trial
Brief Title: Diagnosing Deep-vein Thrombosis Early in Critically Ill Patients
Acronym: DETECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC 20/257/R
Record Dates: First submitted 2021-10-26; First posted 2021-11-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Group (Active Comparator): Patients will be receiving twice weekly proximal lower limb ultrasound
  Interventions: Diagnostic Test: Proximal lower limb ultrasound
- Control Group (No Intervention): Proximal lower limb ultrasound will be performed as per the treating team discretion

INTERVENTIONS:
Diagnostic Test: Proximal lower limb ultrasound — Twice weekly proximal lower limb ultrasound
  Arms: Ultrasound Group

SUMMARY:
The DETECT randomized controlled trial addresses the question of whether surveillance ultrasound in critically ill patients by facilitating DVT detection reduces the incidence of PE and lowers all-cause 90-day mortality. The primary outcome is 90-day all-cause mortality.

DETAILED DESCRIPTION:
This is an open-label multicenter multinational randomized-controlled trial. All patients admitted to ICU will be screened within the first 48 hours of ICU admission for eligibility. Subjects who meet all criteria for enrollment will be randomized via a password-protected, secure website using a variable-size block concealed computer-generated randomization procedure. Patients will be allocated to twice weekly bilateral lower limb ultrasound or standard care (control) in a 1:1 ratio.

ELIGIBILITY:
Inclusion criteria

1. Medical, surgical or trauma ICU patients ≥18 years old.
2. Patients who are expected to stay in the ICU more than 2 calendar days (unlikely to be discharged out of ICU on the day of admission or on the next day).

Exclusion Criteria

1. Patients with DVT or PE diagnosed within the last year.
2. Patients receiving chronic systemic anticoagulation.
3. Patients who have received up to the time of ICU admission or are receiving therapeutic doses of anticoagulation with UFH, LMWH, or other anticoagulants.
4. Inability or contraindication to obtain adequate ultrasound on the lower extremities (Burns in the lower extremities, lacerations, active skin infection, & ischemic limb in the legs, large dressings in the thighs that prevent adequate ultrasounds OR amputated foot or leg on one or two sides)
5. Patients with Inferior Vena Cava (IVC) Filter.
6. Known or suspected pregnancy.
7. Limitation of life support, life expectancy <7 days or palliative care.
8. Previously enrolled in DETECT trial within the last 180 days.
9. Enrolled in another trial for which co-enrolment is not approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | 90 days
  Mortality 90 days post randomization

SECONDARY OUTCOMES:
Proximal DVT | From randomization date to day 28 or ICU discharge whichever comes first
  Lower limb proximal leg DVT, defined as partially or completely incompressible venous segment.
Pulmonary Embolism | From randomization date and throughout hospital stay up to day 28
  Pulmonary embolism defined as definite PE (characteristic intraluminal filling defect on CT chest, high probability VQ scan or detected at autopsy); probable PE (moderate-high pretest, no test or a non-diagnostic test); possible PE (low pre-test probability, non-diagnostic test) or No PE (negative or normal test)
Clinically important bleeding | From randomization date and throughout hospital stay up to day 90
  Fatal bleeding, symptomatic bleeding in critical organ or bleeding causing fall in hemoglobin, requiring transfusion or interventional radiology

OTHER OUTCOMES:
Mechanical ventilation-free days | 28 days
  Total number of days alive and free of mechanical ventilation within 28 days after randomization
Vasopressor-free days | 28 days
  Total number of days alive and free of vasopressor use within 28 days after randomization
Days alive and out of hospital by day 90 | 90 days
  Days alive and out of the hospital at day 90 calculated by using the days from alive at hospital discharge to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Yaseen M Arabi, Principal Investigator — King Saud bin Abdulaziz University of Health Sciences
Locations (1):
- King Abdulaziz Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data supporting this study's findings will be available from the corresponding author upon reasonable request as per the regulations of King Abdullah International Medical Research Center (KAIMRC).
Time Frame: After the publication of the main manuscript (Primary outcome analysis)
Access Criteria: Proposal that describes planned analyses must be submitted along with a data sharing agreement

REFERENCES:
- [Derived] Arabi YM, Alenezi F, Al-Hameed F, Al Humedi HI, Kharaba A, Alhazzani W, Alshahrani MSS, Algethamy H, Maghrabi K, Chalabi J, Ardah HI, Alahmari AM, AlQahtani RM, Ababtain AA, Al-Filfil WAM, Al-Fares AA, Buabbas SF, Bin Humaid F, Brembali MJ, Amer M, Sadat M, Al Tamimi A, AlHumaidan A, Alqahtani M, Al-Dawood A; Saudi Critical Care Trials Group. Diagnosing deep vein thrombosis early in critically ill patients (DETECT) trial: a protocol for a randomised controlled trial. BMJ Open. 2025 Oct 29;15(10):e104468. doi: 10.1136/bmjopen-2025-104468. PMID 41161824